CLINICAL TRIAL: NCT03154515
Title: Randomised Double Blind Placebo Controlled Multicenter Study for Evaluation of Clinical Efficacy and Safety of Ingavirin 90 mg Once Daily to Treat Influenza and Other Acute Viral Infections in Adults.
Brief Title: Efficacy and Safety Study of Ingavirin® 90 mg Once Daily to Treat Influenza and Other Acute Viral Infections in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5P/08
Record Dates: First submitted 2017-04-26; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Common Cold; Influenza, Human; Acute Respiratory Infection
Keywords: Respiratory Tract Infections; Acute Respiratory Viral Infection
MeSH Terms: conditions — Common Cold; Influenza, Human; Respiratory Tract Infections | interventions — pentanedioic acid imidazolyl ethanamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ingavirin (Experimental): Imidazolyl ethanamide pentandioic acid 90 mg once daily for 5 days
  Interventions: Drug: Ingavirin
- Placebo (Placebo Comparator): Placebo capsule identical in appearance to Ingavirin capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ingavirin
  Other Names: Imidazolyl ethanamide pentandioic acid
  Arms: Ingavirin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Ingavirin® 90 mg once daily is effective and safe for the treatment of influenza and other laboratory confirmed acute respiratory viral infections in the course of standard therapy in patients 18-60 years old.

DETAILED DESCRIPTION:
Randomized, Multicenter, Double-Blind, Parallel-Group, Placebo-Controlled Trial of the Efficacy and Safety of Ingavirin in the Treatment of Influenza and Other Acute Viral Respiratory Infection. Study treatment was 5 days followed by 2 ± 1 days of follow up period. Thus, study participation was 7 ± 1 days (8 days max).

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically diagnosed influenza, body temperature ≥ 38 ºС or other acute respiratory viral infection, body temperature ≥ 37 ºС, with no less than 2 symptoms of catarrhal and intoxication each:

  * Intoxication symptoms: Dizziness, headache, chills, fever, sweating, fatigue, myalgia, pain while moving eyes, flushing, pale skin, sleep disturbances, decreased appetite, nausea, vomiting, epistaxis, cyanosis, meningeal signs.
  * Catarrhal symptoms: Sore throat, rhinorrhea and nasal congestion, difficulty swallowing, hoarseness, stridor, wheezing, rattling dry and wet cough, expectoration.
* Laboratory confirmation of viral origin of the disease
* Uncomplicated influenza and other acute respiratory viral infections
* Interval between onset of symptoms and enrollment to the study not more than 48 hours
* Have read, understood and signed an informed consent form

Exclusion Criteria:

* Complicated course of influenza and other acute respiratory viral infections (secondary bacterial infection)
* Pregnancy and Breastfeeding
* Severe decompensated or unstable medical or psychiatric conditions (any diseases or conditions that threaten the life of the patient or worsen the patient's prognosis)
* Cancer, HIV infection, tuberculosis, including those in history
* History of alcohol and drug abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 445 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Time to resolution of fever | 7 ± 1 days
  Time from the start of study treatment to resolution of fever ( t ≤ 36,9 ºС, till the end of the follow up).

SECONDARY OUTCOMES:
Time to resolution / alleviation of intoxication symptoms | 7 ± 1 days
  Following symptoms were recorded and rated each visit, to evaluate symptoms progress:
  Dizziness, headache, chills, fever, sweating, fatigue, myalgia, pain while moving eyes, flushing, pale skin, sleep disturbances, decreased appetite, nausea, vomiting, epistaxis, cyanosis, meningeal signs.
Time to resolution / alleviation of catarrhal symptoms | 7 ± 1 days
  Following symptoms were recorded and rated each visit, to evaluate symptoms progress:
  Sore throat, rhinorrhea and nasal congestion, difficulty swallowing, hoarseness, stridor, wheezing, rattling dry and wet cough, expectoration.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Through study completion, an average of 8 days
  All adverse events recorded and analysed, to compare incidence rate with one of placebo.
  Complete blood count test performed at the beginning and at the end of the study.
  Vital signs taken and recorded at each visit throughout the study, usually every day for 7 ± 1 days.

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Zakharova, MD, PhD, Study Director — Valenta Pharm JSC
Locations (9):
- Russia (9):
  - State educational institution of higher professional education "Chelyabinsk State Medical Academy of Federal Agency of Health Care and Social Development", Chelyabinsk
  - N.F. Gamaleya Scientific Research Institute of Epidemiology and Microbiology, Moscow
  - State budgetary health care institution novosibirsk region "city clinical infectious diseases hospital no. 1", Novosibirsk
  - North-western State Medical University named after I.I.Mechnikov, Saint Petersburg
  - Saratov State Medical University named after V. I. Razumovsky, Saratov
  - Federal State Budgetary Educational Institution of Higher Education "Pacific State Medical University" of the Ministry of Healthcare of the Russian Federation, Vladivostok
  - Volgograd State Medical University, Volgograd
  - Yaroslavl State Medical University, Yaroslavl
  - Federal State Budgetary Institution of Higher Professional Education "Urals State Medical University" of the Ministry of Healthcare of the Russian Federation, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No